CLINICAL TRIAL: NCT03066427
Title: Phase II Study to Evaluate Efficacy and Safety of Sunitinib Therapy in Patients With Metastatic Renal Clear Cell Carcinoma Who Have Progressed to First-line Immunotherapy Treatment (INMUNOSUN Study)
Brief Title: Study to Evaluate Efficacy and Safety of Sunitinib in Renal Cell Carcinoma Progressed to 1L Immunotherapy Treatment.
Acronym: INMUNOSUN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Spanish Oncology Genito-Urinary Group (Other)
Collaborators: Pfizer (Industry); Apices Soluciones S.L. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SOGUG-2016-A- IEC(REN)-10; 2016-004011-12 (EudraCT Number)
Record Dates: First submitted 2017-02-23; First posted 2017-02-28 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-10

CONDITIONS: Clear Cell Renal Carcinoma
Keywords: Clear Cell Renal Carcinoma; Sunitinib
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sunitinib (Experimental): Sunitinib 50 mg/day, 4 weeks on/2weeks off
  Interventions: Drug: Sunitinib

INTERVENTIONS:
Drug: Sunitinib — Sunitinib 50 mg/d
  Other Names: Sutent

SUMMARY:
The therapeutic scenario of metastatic renal cancer is undergoing a new revolution with the appearance of a novel therapeutic strategy after the antiangiogenic treatments, that is the immunotherapy, in addition to the approval of new active drugs in the following lines of treatment.

There are currently two phase III trials in the first line of treatment in metastatic renal cancer that include different combinations of treatment based on immunotherapy. If results of these studies were positive, the therapeutic algorithm would be modified so that the remaining drugs would have to be repositioned within the therapeutic decision scheme.

Sunitinib has previously demonstrated its benefit in patients who had failed to prior treatment with cytokines, so it is likely to continue to be effective in patients who have become resistant to treatment with new drugs based on immune checkpoint blockade.

This phase II study is developed to evaluate the activity of sunitinib after treatment with immunotherapy-based regimens that are currently being developed within phase III clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* 1. Eighteen years or older on the day of consent
* 2. Documented histological or cytological diagnosis of renal cell cancer with a clear-cell component.
* 3. Patient must have progressed to at least one immune check point inhibitor-based therapy (antiPD1, anti-PDL1 o antiCTLA4) for the first line
* 4. Measurable disease per RECIST 1.1 as determined by the investigator
* 5. The subjects should not present disease that may be subsidiary of surgical treatment, radiotherapy or combined treatment with curative intent.
* 6. Recovery of toxicities related to any prior treatments to ≤ Grade 1 CTCAE v.4.03, unless adverse event(s) are clinically nonsignificant and/or stable on supportive therapy.
* 7. Eastern Cooperative Oncology Group Performance Status (PS) 0-2
* 8. Adequately controlled blood pressure (BP) with or without antihypertensive medication to maintain a BP <150/90 mmHg before the start of study treatment.
* 9. Adequate marrow function

  * Absolute neutrophil count (ANC) ≥ 1500/mm3 (≥ 1.5 GI/L).
  * Platelets ≥ 100,000/mm3 (≥ 100 GI/L).
  * Hemoglobin ≥ 9 g/dL (≥ 5,6 mmol/L).
* 10. Adequate liver function

  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 2.5 × ULN.
  * Total bilirubin ≤ 1.5 × upper limit of normal (ULN).
* 11. Adequate kidney function: calculated creatinine clearance ≥ 30 mL/min (≥ 0.5 mL/sec) using the Cockroft-Gault equation
* 12. Proteinuria <2+ on urine test strip
* 13. Prothrombin Time (PT) or International Standard Ratio (INR) ≤ 1.2 x ULN.
* 14. Life expectancy >3 months.
* 15. Patient able to ingest study drug and meet study follow-up requirements.
* 16. Sexually active fertile subjects and their partners must agree to use medically accepted methods of contraception
* 17. Female subjects of childbearing potential must not be pregnant at screening.

Exclusion Criteria:

* 1. Previous treatments with sunitinib are not permitted for the advanced or localized disease.
* 2. Major surgery within 3 weeks of patient inclusion
* 3. Radiation therapy or embolization within 2 weeks of first dose of sunitinib
* 4. Previous treatment with immunosuppressive drugs such as cyclosporine, tacrolimus, azathioprine, or long-term oral glucocorticoids taken prior to (3 months) patient inclusion
* 5. Prior high-dose chemotherapy requiring hematopoietic stem cell rescue.
* 6. Current treatment on another clinical trial.
* 7. Treatment with known potent CYP3A4 inhibitors or inducers or that prolong the QT interval, within 7 days prior to the inclusion.
* 8. Prior radiation therapy to >25% of the bone marrow.
* 9. Uncontrolled brain metastases, spinal cord compression, carcinomatous meningitis, or leptomeningeal disease.
* 10. Any gastrointestinal malabsorption disorder or any other condition that, in the opinion of the investigator, may affect the absorption of sunitinib or increase the risk of bleeding or perforation.
* 11. Presence of an unhealed wound or active ulcer.
* 12. Diarrhea grade III/IV in the screening period.
* 13. Diagnosis of any second malignancy within the last 3 years, except for adequately treated basal cell or squamous cell skin cancer, or carcinoma in situ of the cervix.
* 14. Clinically significant cardio-cerebrovascular disease within 6 months prior to initiation of treatment.
* 15. Ongoing cardiac dysrhythmias of NCI CTCAE grade ≥2, atrial fibrillation of any grade that require treatment.
* 16. Corrected QT interval (QTc) interval >500 msec.
* 17. Active hemoptysis within 6 weeks prior to initiation of study treatment.
* 18. Evidence of active bleeding or hemorrhagic diathesis.
* 19. Presence of endobronchial lesions and / or lesions that infiltrate large vessels.
* 20. Current treatment with therapeutic doses of Coumadin (low dose Coumadin up to 2 mg PO daily for deep vein thrombosis prophylaxis is allowed).
* 21. Other clinically significant alterations:

  * Known human immunodeficiency virus (HIV) infection.
  * Presence of an uncontrolled active infection.
  * Presence of uncontrolled or symptomatic hypothyroidism.
  * Moderate-severe liver disease (Child Pugh B-C).
  * Requirement for hemodialysis or peritoneal dialysis.
  * History of solid organ transplantation.
* 22. Pregnancy or breastfeeding.
* 23. Any disease that, in the opinion of the investigator, interferes with the patient's ability to participate in the clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2017-05-10 (Actual); Primary Completion 2020-09-22 (Actual); Study Completion 2020-09-22 (Actual)

PRIMARY OUTCOMES:
Objective response rate | 12 months
  Percentage of patients with documented response according RECIST 1.1 criteria (complete response + partial response)

SECONDARY OUTCOMES:
Progression-free survival | 12 months
  Time from start of treatment to disease progression or death.
Time to progression | 12 months
  Time from start of treatment to disease progression or death due to the illness
Duration of the response | 12 months
  Time from first response to disease progression or death.
Overall survival | 18 months
  Time from start of treatment to death.
Clinical benefit | 12 months
  Percentage of patients with documented response or disease stabilization according RECIST 1.1 criteria
Number of individual events (hematologic events and not hematologic events) | 12 months
  Percentage of patients with each of the adverse event per grade

CONTACTS AND LOCATIONS:
Overall Officials: Enrique Grande, MD, Study Chair — MD Anderson Cancer Center Madrid; Cristina Suárez, MD, Principal Investigator — Hospital Vall d'Hebron; Xavier García del Muro, MD, Principal Investigator — Hestia Duran i Reynals; Oscar Reig, MD, Principal Investigator — Hospital Clínic i Provincial de Barcelona; María J Méndez, MD, Principal Investigator — Complejo Hospitalario Regional Reina Sofia; Daniel Castellano, MD, Principal Investigator — Hospital Universitario 12 de Octubre; Teresa Alonso, MD, Principal Investigator — Hospital Universitario Ramon y Cajal
Locations (9):
- Spain (9):
  - ICO Duran i Reynals, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clínic i Provincial de Barcelona, Barcelona
  - Complejo Hospitalario Regional Reina Sofía, Córdoba
  - Hospital Ramón Y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Centro Integral Oncologico Clara Campal, Madrid
  - MD Anderson Cancer Center Madrid, Madrid
  - Hospital Central de Asturias, Oviedo

IPD SHARING:
Plan to Share IPD: No